CLINICAL TRIAL: NCT04401410
Title: BAT IT: Banked Anti-SARS Cov-2 T Cell Infusions for Treatment of COVID 19
Brief Title: Anti-SARS Cov-2 T Cell Infusions for COVID 19
Acronym: BATIT
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to trial's eligibility criteria and the low census of hospitalized COVID-19 patients meeting eligibility criteria, the Sponsor will be unable to enroll a meaningful number of patients in this single-center trial in a reasonable time frame.
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other); AlloVir (Industry); The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Premal Lulla, Assistant Professor, Baylor College of Medicine
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-47739 BAT IT
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: SARS-CoV 2; Viral Infection; COVID 19
Keywords: COVID 19; SARS-CoV 2; Viral infection; Multivirus T cell
MeSH Terms: conditions — Virus Diseases; COVID-19 | interventions — Maximum Tolerated Dose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dose Finding Phase (Experimental): This phase is designed to evaluate the maximum tolerated dose (MTD) of partially HLA-matched SARS-CoVSTs administered to hospitalized COVID19 patients with high risk of progression to mechanical ventilation.
  The dose finding phase is a standard 3+3 safety study design. The 3 dose levels are:
  DL1: 1x10^7 cells (flat dose) DL2: 2x10^7 cells (flat dose) DL3: 4x10^7 cells (flat dose)
  Interventions: Biological: Dose Finding Phase (MTD)
- Randomized Pilot - SARS-CoVSTs (Experimental): Partially HLA-matched Virus Specific T cells (VSTs) will be given by intravenous injection.
  Interventions: Biological: Partially HLA-matched SARS-CoVSTs
- Randomized Pilot - Routine Care (Active Comparator): Hospitalized patients with COVID-19 will be treated per current institutional guidelines.
  Interventions: Other: Routine care (no SARS-CoVSTs)

INTERVENTIONS:
Biological: Dose Finding Phase (MTD) — Enrollment to the dose escalation phase will be staggered. The first patient enrolled on each of the 3 dose levels (DL1, DL2 and DL3) will have to complete the 14-day toxicity monitoring window prior to enrollment of the next patients. Prior to dose escalation, all patients at a particular dose level should have completed the minimum 14-day toxicity monitoring window before enrolling to a higher dose level.
  Arms: Dose Finding Phase
Biological: Partially HLA-matched SARS-CoVSTs — Infusion of SARS-CoVSTs at the MTD level as determined in the Dose Finding Phase
  Arms: Randomized Pilot - SARS-CoVSTs
Other: Routine care (no SARS-CoVSTs) — Patients receive routine care for COVID19 per institutional standards (including antivirals such as remdesivir or other FDA-EUA approved products and thromboprophylaxis).
  Arms: Randomized Pilot - Routine Care

SUMMARY:
This is a dose-finding safety trial followed by a randomized pilot trial comparing administration of SARS-CoV2-specific T cells (SARS-CoVSTs) to standard of care treatment in hospitalized patients with COVID19 who are at high risk of requiring mechanical ventilation.

The SARS-CoVSTs lines have been made at Baylor College of Medicine from healthy donors who have made a full recovery from COVID19. These cell lines were frozen for later use and will be thawed and used to treat patients who meet the eligibility criteria.

DETAILED DESCRIPTION:
The first part of this study is to identify the maximum tolerated dose (MTD) of allogeneic SARS-CoV2-specific T cells (SARS-CoVSTs) for patients with COVID19 with high risk of progression to mechanical ventilation.

The 3 dose levels (DL) are:

DL1: 1x10^7 cells (flat dose) DL2: 2x10^7 cells (flat dose) DL3: 4x10^7 cells (flat dose)

Enrollment to the dose escalation phase will be staggered. The first patient enrolled on each of the 3 dose levels (DL1, DL2 and DL3) will have to complete the 14-day toxicity monitoring window prior to enrollment of the next patients. Prior to dose escalation, all patients at a particular dose level should have completed the minimum 14-day toxicity monitoring window before enrolling to a higher dose level.

After the dose finding phase is complete and the MTD established, a randomized trial will be conducted. Patient will be randomized 1:1 using the permuted block method with a block size of 4 (2 in the treatment arm and 2 in the control arm) to receive treatment with SARS-CoVSTs or routine treatment per institutional standards.

All enrolled patients will undergo the following evaluations:

* Physical exam and history including height and weight
* SARS-CoV-2 test
* Blood tests
* Chest X-ray or chest CT Scan if not already done in the past 48 hours.
* A urine pregnancy test, when applicable

Patients randomized to receive SARS-CoVSTs will be pre-medicated with Benadryl and Tylenol. The cells will be thawed and given through an intravenous line. Patients will be monitored for infusion side effects for up to 14 days or until infusion side effects have completely resolved, whichever is longer.

Blood will be drawn before the infusion and then up to daily for 14 days or until the patient is discharged from the hospital. Optional blood samples will be drawn at 2, 3 and 6 months after infusion. Study participation will last 6 months after the date of infusion.

ELIGIBILITY:
Inclusion Criteria

1. SARS-CoV-2 infection confirmed by polymerase chain reaction assay (PCR) from a nasopharyngeal swab or other accepted specimen type. (If testing was performed ≥ 5 days before enrollment, this must be repeated and accept only if positive again). Date of COVID test must be ≤ 5 days prior to infusion.
2. Currently hospitalized adult patient (≥ 18 years of age) requiring medical care for COVID19
3. Peripheral oxygen saturation (SpO2) ≥ 92% on room air
4. Hgb ≥ 7.0 gm/dl
5. Negative pregnancy test (if applicable)
6. Patient or parent/guardian capable of providing informed consent (may be obtained electronically)
7. Evidence of pulmonary infiltrates on chest imaging. Any chest imaging findings which would be consistent with COVID19 would qualify (Eg: ground glass opacities, multifocal infiltrates etc.)
8. High risk of requiring mechanical ventilation as defined by at least two of the following:

   1. Age ≥ 60 years of age
   2. Age ≥ 75 years of age (counts as meeting two criteria)
   3. Hypertension (HTN)
   4. Chronic cardiovascular disease other than HTN (eg: Coronary artery disease, congestive heart failure or cardiomyopathies).
   5. Diabetes Mellitus
   6. Obesity (BMI ≥ 30)
   7. Obesity (BMI ≥ 40, counts as meeting two criteria)
   8. Active cancer diagnosis or ongoing (within 3 months) cytotoxic chemo/ radio-therapy for a cancer
   9. Post-hematopoeitic stem cell or solid organ transplantation status
   10. Immunodeficiency states including HIV infection on antiretroviral therapy (except those listed as exclusion criteria #1, #7 and #10) as determined by the treating physician (eg: receiving immunosuppressive therapy like rituximab or congenital immunodeficiency syndromes, prior treatment with chemotherapy greater than 3 months ago but per investigators discretion could have lingering effects on the immune system, eg: chemotherapy regimens for lymphomas, ALL or AML etc.)
   11. Chronic obstructive pulmonary disease (COPD)
   12. Current everyday smoker
   13. Chronic kidney disease (eGFR < 30 mL/min/1.73 m2 )
   14. Bronchial asthma (on active treatment prior to admission, eg. Use of rescue inhalers or inhaled corticosteroids or other treatments to prevent/treat attacks).

Exclusion Criteria

1. Received Anti-thymocyte globulin (ATG), Campath or other T cell immunosuppressive monoclonal antibodies in the 28 days prior to screening for enrollment
2. Requiring mechanical ventilation at time of T cell infusion
3. Alanine aminotransferase or aspartate aminotransferase greater than 5 x upper limit of normal
4. If previously undergone an allogeneic hematopoietic stem cell transplant and have evidence of active acute GVHD greater than or equal to grade 2
5. Uncontrolled relapse of malignancy
6. Requiring vasopressors
7. Known history of autoimmune disease except prior thyroiditis
8. Is not suitable at the discretion of the treating physician
9. Patients on greater than 6mg/day of dexamethasone (IV) or equivalent
10. Greater than grade 1 CRS per American Society for Transplantation and Cellular Therapy (ASTCT) criteria
11. Patients should not be enrolled on any other interventional clinical trials for COVID19. Patients may receive routine care for COVID19 per institutional standards (including antivirals such as remdesivir or other FDA-EUA approved products and thromboprophylaxis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-10-12 (Actual)

PRIMARY OUTCOMES:
Dose Escalation Phase: Rate of Dose Limiting Toxicities by CTCAE 5.0 [14 days post infusion] | 14 days post infusion
  Defined as the proportion of subjects with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment. A dose limiting toxicity is defined as any acute GvHD (> grade 2), grade ≥3 CRS or ICANS, grade ≥3 hematologic toxicity or grade ≥3 non-hematologic adverse events related to the T cell product within 14 days of the VST infusion and that are not due to pre-existing conditions as defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.
Randomized Trial: Rate of Clinical Response as assessed by the World Health Organization (WHO) Ordinal Scale [7 days post-randomization or hospital discharge] | 7 Days post-randomization or at time of hospital discharge
  Clinical Response rate is defined as the proportion of subjects reporting an increase in 2 or more points on the WHO Ordinal Scale. [Scored on a scale from 0 to 8; where 0 = Uninfected and 8 =Dead] or until patient is discharged.

SECONDARY OUTCOMES:
Randomized Trial: Rate of Treatment-related adverse events (tAE) by CTCAE 5.0 [14 days post-randomization] | 14 days post-randomization
  Defined as the proportion of subjects with toxicity including the type, severity, time of onset, time of resolution, and the probable association with study treatment. Treatment-related adverse events (tAE) are defined as any acute GvHD (> grade 2), grade ≥3 CRS or ICANS, grade ≥3 hematologic toxicity or grade ≥3 non-hematologic adverse events related to the T cell product within 14 days of the VST infusion and that are not due to pre-existing conditions as defined by the NCI Common Terminology Criteria for Adverse Events (CTCAE), Version 5.

CONTACTS AND LOCATIONS:
Overall Officials: Premal Lulla, Principal Investigator — Baylor College of Medicine
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

REFERENCES:
- [Derived] Vasileiou S, Hill L, Kuvalekar M, Workineh AG, Watanabe A, Velazquez Y, Lulla S, Mooney K, Lapteva N, Grilley BJ, Heslop HE, Rooney CM, Brenner MK, Eagar TN, Carrum G, Grimes KA, Leen AM, Lulla P. Allogeneic, off-the-shelf, SARS-CoV-2-specific T cells (ALVR109) for the treatment of COVID-19 in high-risk patients. Haematologica. 2023 Jul 1;108(7):1840-1850. doi: 10.3324/haematol.2022.281946. PMID 36373249

DOCUMENTS (1):
  • Informed Consent Form (2020-09-28): https://cdn.clinicaltrials.gov/large-docs/10/NCT04401410/ICF_000.pdf